CLINICAL TRIAL: NCT05112497
Title: Mother-to-Infant Transfer of Bacteriome, Fungome, Virome, and Metabolome in Health and Crohn's Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: First Affiliated Hospital of Kunming Medical University (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: MoMmy-CD
Record Dates: First submitted 2021-05-05; First posted 2021-11-09 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Gut Microbiota; Mother-baby Cohort
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's Disease: 1. Pregnant CD patients
  2. Newborn of pregnant CD patients
  3. Father of the newborn
  4. Non-pregnant CD women
  Interventions: Other: No intervention procedure
- Healthy Control: 1. Pregnant women without CD
  2. Newborn of pregnant women without CD
  3. Father of the newborn
  Interventions: Other: No intervention procedure

INTERVENTIONS:
Other: No intervention procedure — No intervention procedure

SUMMARY:
Inflammatory bowel diseases (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), are caused by the loss of mucosal tolerance towards the commensal microbiota resulting in inflammatory responses. Both CD and UC are difficult to manage clinically, and their incidences are increasing worldwide especially in newly industrialized countries. The etiology of these disorders is multifactorial, influenced by the complex interactions of genes, the immune system, intestinal microbiota, and the external environment. Studies have shown that there is a higher disease transmission rate from mothers with IBD than from fathers. It is well established that IBD is also associated with perturbations of gut microbiota composition. Early childhood is a golden age for microbiota manipulation to prevent disease. Studying microbiota at this golden age also allow us to dissect the development of a faulty microbiota and identify therapeutic targets to reverse it and cure diseases that are already developed. New evidence suggests that the gastrointestinal tract of new-borns becomes colonized with bacteria while in the womb, with the presence of different microbes. The source of these microbes is of continued interest because the initial intestinal colonization is believed to play a crucial role in the priming of the mucosal immune system and may predispose to the development of immune-mediated diseases, such as IBD, later in life. Overall, the microbiome structures in mother-babies across healthy and IBD populations are largely underexplored.

Given the complexity of microbes present in the gestational gut, it will be exciting to learn whether there are other modules of priming induced by distinct microbes and their metabolites. Along these lines, it is tempting to speculate that this transgenerational effect represents a predictive adaptive response whereby mothers prepare the neonates for specific challenges that they are likely to encounter based on gestational environmental cues, not only by microbial colonisation but also by metabolite transfer. Meanwhile, it is unknown whether there are abnormalities in the metabolome and its mother-to-infant transfer in IBD. Those results indicate that the metabolomic profiles are altered in IBD mother's breast milk, which may transfer to infants and influence their development and health.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), are caused by the loss of mucosal tolerance towards the commensal microbiota resulting in inflammatory responses. Both CD and UC are difficult to manage clinically, and their incidences are increasing worldwide especially in newly industrialized countries. The etiology of these disorders is multifactorial, influenced by the complex interactions of genes, the immune system, intestinal microbiota, and the external environment. Studies have shown that there is a higher disease transmission rate from mothers with IBD than from fathers.[47] It is well established that IBD is also associated with perturbations of gut microbiota composition. Early childhood, when the microbiota is less mature and more malleable, is a golden age for microbiota manipulation to prevent disease. Studying microbiota at this golden age also allow us to dissect the development of a faulty microbiota and identify therapeutic targets to reverse it and cure diseases that are already developed. New evidence suggests that the gastrointestinal tract of new-borns becomes colonized with bacteria while in the womb[1], with the presence of different microbes reported in amniotic fluid[2, 3], umbilical cord blood[4], as well as placental and foetal membranes[5, 6]. The source of these microbes is of continued interest because the initial intestinal colonization is believed to play a crucial role in the priming of the mucosal immune system and may predispose to the development of immune-mediated diseases, such as IBD, later in life[7]. Our pilot study on several mother-baby samples showed that at the order level, Caudovirales predominated in the viral communities of breast milk and meconium with relative abundance above 95%. However, in the viral community of placenta, the Caudovirales only occupied approximately 50%, concomitant with the emergence of eukaryotic viruses such as Ortervirles (average 27.5%) and Herpesvirales (average 9.3%). Overall, the microbiome structures in mother-babies across healthy and IBD populations are largely underexplored.

A recent study discovered a novel mechanism of vertically transmitted protection of the new-born. The researchers found that bacteria in the mother's intestine during gestation can drive later innate maturation of the neonatal gut in the absence of colonization, through the transfer of specific bacterial metabolites to the foetus and via mother's milk [8]. Gomez de Agu ero et al. (2016) clearly demonstrated that the effects of the gut microbiota on postnatal immune maturation are not simply due to colonization of the new-born after birth[9]. They show this in a simplified model of gestational monocolonization with E. coli whereby AhR ligands derived from this bacterium drive a distinct early postnatal intestinal developmental program[9]. Given the complexity of microbes present in the gestational gut, it will be exciting to learn whether there are other modules of priming induced by distinct microbes and their metabolites. Along these lines, it is tempting to speculate that this transgenerational effect represents a predictive adaptive response whereby mothers prepare the neonates for specific challenges that they are likely to encounter based on gestational environmental cues, not only by microbial colonisation but also by metabolite transfer. Meanwhile, it is unknown regarding whether there are abnormalities in the metabolome as well as its mother-to-infant transfer in IBD. To address this question, we began with a pilot study on breast milk metablome profiling, employing untargeted metabolomics approach by liquid chromatography-mass spectrometry (LC-MS). The results showed a total of 1,318 Negative-mode features and 1,418 Positive features discriminatory between IBD (4UC, 3 CD) mothers and healthy mothers, indicative of broad metabolic differences between them. Those significantly changed metabolites were involved in arginine and proline metabolism as well as tyrosine metabolism according to pathway enrichment analysis. Those results indicate that the metabolomic profiles are altered in IBD mother's breast milk, which may transfer to infants and influence their development and health.

ELIGIBILITY:
Inclusion Criteria for CD patients:

* To be pregnant in the 1st trimester or planning pregnancy.
* Diagnosis of Crohn's disease is confirmed by clinical, endoscopic, radiological and histological features
* All eligible should sign the consent form

Inclusion Criteria for Healthy Control:

* To be pregnant in the 1st trimester or planning pregnancy
* Subjects without a diagnosis of IBD
* All eligible should sign the consent form

Inclusion Criteria for non-pregnant CD patients

* Diagnosis of Crohn's disease is confirmed by clinical, endoscopic, radiological and histological features
* All eligible should sign the consent form

Exclusion Criteria for all groups:

* Co-morbidities, such as type I or type II diabetes, autoimmune diseases, cancer, HIV
* Inability to give informed consent
* Probiotics. prebiotics and antibiotics use in the past 3 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CD:
  1. Pregnant CD patient
  2. Newborn of pregnant CD patient
  3. Father of newborn
  4. Non-pregnant CD women
  Healthy:
  1. Pregnant women without CD
  2. Newborn of pregnant women without CD
  3. Father of newborn
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
The gut metagenomes at the bacteria species level the among different groups will be determined | across two years
  Metagenomic sequencing will be used to evaluate the heterogeneities of the bacteria species among different groups.

SECONDARY OUTCOMES:
The temporal dynamics of the development of the breast milk microbiota in mothers and infants will be determined | across two years
  Metagenomic sequencing will be used to evaluate the heterogeneities of the bacteria species of breast milk in mothers and infants.

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No